CLINICAL TRIAL: NCT02372318
Title: Nalmefene Challenge to Modulate Neural Reactivity to Alcohol-related and Emotional Cues in Non-treatment Seeking Alcohol Dependent Participants
Brief Title: Single-dose of Nalmefene to Modulate Neural Alcohol Cue Reactivity
Acronym: NALCUE
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Anticipated nr of 25 probands was not reached in terms of full data sets (missing data, low fMRI data quality), but time frame for recruitment ended.
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Lundbeck GmbH, Ericusspitze 2, 20457 Hamburg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 37
Record Dates: First submitted 2015-02-06; First posted 2015-02-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-01

CONDITIONS: Alcoholism
Keywords: opiod receptor modulator nalmefene; cue-reactivity; fMRI; resting-state networks
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nalmefene Challenge (Experimental): Participants will receive 18mg Nalmefene two hours prior to fMRI measurement. During fMRI scanning alcohol cues will be presented.
  Interventions: Drug: Nalmefene
- Placebo (Placebo Comparator): Participants will receive Placebo two hours prior to fMRI measurement. During fMRI scanning alcohol cues will be presented.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalmefene — 18mg of Nalmefen will be administered orally
  Other Names: Selincro
  Arms: Nalmefene Challenge
Drug: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The aim of this study is to use functional Magnetic Resonance Imaging (fMRI) to measure neural reactivity to alcohol-related and emotional cues in alcohol dependent subjects following a single dose of the opioid receptor modulator nalmefene. The study will be done in a cross over design with nalmefene versus placebo.

DETAILED DESCRIPTION:
All subjects will undergo a battery of minimal risk procedures during each study visit; filling out questionnaires, performing agreed behavioral tasks, scanning procedures including two functional MRI (fMRI) scans as well as structural MRI.

The fMRI will be obtained in non-abstinent participants with breath alcohol concentrations not larger than > 0.3 ‰ and withdrawal severity not more than 4 on the clinical institute withdrawal assessment for alcohol (CIWA-Ar) scale.

Alcohol consumption will be assessed with the Form90 interview. Severity of alcohol dependence will be examined with the Alcohol Dependence Scale (ADS). Drinking situations will be assessed with the Inventory of Drinking Situations (IDS). Trait aspects of craving for alcohol will be measured with the Obsessive Compulsive Drinking Scale (OCDS). To examine state and trait anxiety the State-Trait Anxiety Inventory (STAI) will be used. Depressive symptoms will be measured with the Beck Depression Inventory (BDI) and the State-Trait Depression Scales (STDS). Nicotine consumption will be assessed with the Fagerström Test for Nicotine Dependence.

The following scales will be administered before and after each fMRI scanning: The Alcohol Craving Questionnaire (ACQ), the Alcohol Urge Questionaire (AUQ) and visual analogue scales for craving assessment.

Participants will undergo two fMRI scanning sessions at intervals of one week: one 2 h after administration of nalmefene and one 2 h after administration of placebo, carried out in a randomized order.

MRI examinations include

* a cue-reactivity task;
* an emotional faces task;
* resting-state fMRI;
* structural MRI;
* including preparation, instructions and breaks

ELIGIBILITY:
Inclusion Criteria:

* severe alcohol use disorder according to DSM 5 and "heavy drinking": alcohol consumption >=60g (men) and >=40g (women) (minimum of 5 days / week)
* right-handedness
* normal or corrected to normal vision
* signed written informed consent

Exclusion Criteria:

valid at the time of MRI investigation:

* psychotropic medication within the last 14 days
* severe withdrawal symptoms (CIWA-Ar > 4; Sullivan et al. 1989)
* intoxication (breath alcohol concentration > 0.3 ‰)
* common exclusion criteria for MRI (e.g. metal, claustrophobia)
* positive drug screening (opioids, cannabinoids, benzodiazepines, barbiturates, cocaine, amphetamines)
* pregnancy
* contraindications to the prescription of nalmefene valid at inclusion:
* previous severe withdrawal / withdrawal complications
* previous inpatient detoxification treatment
* other Axis I psychiatric diagnoses than alcohol- or nicotine-dependence in the last 12 months
* neurological disorders, history of brain injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference in cue-induced brain activation between two fMRI scans (randomization to an intake of nalmefene (18 mg) or placebo). | Primary outcome measures will be assessed on day 2 and day3 after fMRI scan, data collection will take up to 12 months
  This difference will be extracted from whole-brain contrast images in the VS and DS using the percentage of activated voxels in these regions of interest (ROI).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim; Falk Kiefer, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Zentralinstitut für Seelische Gesundheit, Mannheim, Germany

REFERENCES:
- [Derived] Grundinger N, Gerhardt S, Karl D, Mann K, Kiefer F, Vollstadt-Klein S. The effects of nalmefene on the impulsive and reflective system in alcohol use disorder: A resting-state fMRI study. Psychopharmacology (Berl). 2022 Aug;239(8):2471-2489. doi: 10.1007/s00213-022-06137-1. Epub 2022 Apr 15. PMID 35426492